CLINICAL TRIAL: NCT05888129
Title: Clinical Outcomes of Surgery After Neoadjuvant Chemotherapy in Locally Advanced Pancreatic Ductal Adenocarcinoma: is it Really Comparable to Borderline Resectable or Resectable Pancreatic Adenocarcinoma?
Brief Title: Clinical Outcomes of Surgery After Neoadjuvant Chemotherapy in Locally Advanced Pancreatic Cancer
Acronym: COSNALAP
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Song Cheol Kim, Professor, Asan Medical Center
Other Study IDs: 2016-0902
Record Dates: First submitted 2023-05-09; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- locally advanced pancreatic cancer: Locally advanced pancreatic cancer (LA-PC) is classified according to the National Comprehansive Cancer Networks (NCCN) guidelines.
  Patients with the above conditions underwent surgery after neoadjuvant chemotherapy.
  Interventions: Procedure: surgery after neoadjuvant chemotherapy
- borderline resectable pancreatic cancer: Borderline resectable pancreatic cancer (BR-PC) is classified according to the NCCN guidelines.
  Patients with the above conditions underwent surgery after neoadjuvant chemotherapy.
  Interventions: Procedure: surgery after neoadjuvant chemotherapy
- resectable pancreatic cancer: Resectable pancreatic cancer (PC) is classified according to the NCCN guidelines.
  There are no arterial and venous contact with tumor Patients with the above conditions underwent upfront surgery

INTERVENTIONS:
Procedure: surgery after neoadjuvant chemotherapy — surgery after neoadjuvant chemotherapy
  Groups: borderline resectable pancreatic cancer; locally advanced pancreatic cancer

SUMMARY:
The purpose of this study was to investigate the clinical outcomes of patients with locally advanced pancreatic cancer (LA-PC) who underwent surgery after neoadjuvant chemotherapy (NACT) at Asan Medical Center's Department of Hepato-Biliary-Pancreatic Surgery from 2017 to 2020.

DETAILED DESCRIPTION:
Pancreatic cancer (PC) has a very low survival rate. Most PC patients have non-specific symptoms that are advanced enough to be contraindications for surgical treatment; therefore, surgery is often impossible by the time PC is diagnosed. According to the NCCN guidelines, PCs with no metastases can be divided into resectable, borderline resectable , and locally advanced cases. Patients with borderline resectable PC (BR-PC) and locally advanced PC (LA-PC) currently receive multimodal therapy before surgery. The goal of these neoadjuvant treatments, including chemotherapy and radiation therapy, is to ultimately reduce local recurrence after surgery in patients with BR-PC and further improve their survival time. Additionally, several recent studies have reported results on the prognosis when surgery is performed after neoadjuvant chemotherapy (NACT) in patients with LA-PC. In the patients with LA-PC, surgery technically difficult because of major vascular invasion before NACT. Therefore, this study investigated the clinical outcomes of patients with LA-PC who underwent surgery after NACT. Additionally, the investigators evaluated factors affecting the prognosis related to survival after surgery in patients with LA-PC.

ELIGIBILITY:
Inclusion Criteria:

* The study population consists of patients who underwent pancreatectomy for pancreatic adenocarcinoma between January 2017 and December 2020

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We retrospectively reviewed records of patients who were diagnosed with resectable, borderline resectable, or locally advanced pancreatic adenocarcinoma between January 2017 and December 2020, at the Department of Surgery, Asan Medical Center, Seoul, South Korea. A total of 1,358 patients were diagnosed with pancreatic ductal adenocarcinoma and treated.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
oncologic outcome | 3 - 5 years after surgery
  overall survival and recurrence free survival according to the groups

CONTACTS AND LOCATIONS:
Overall Officials: Song Cheol Kim, MD. PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No